CLINICAL TRIAL: NCT02635243
Title: SAR438544 - Clinical & Exploratory Pharmacology
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of a Single Dose of SAR438544 in Comparison to Glucagon in Type 1 Diabetes Mellitus Patients Under Induced Hypoglycemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PDY14452; U1111-1172-1152 (Other: UTN)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR438544 dose 1 (Experimental): Single dose of SAR438544 given SC under fasting conditions and under induced hypoglycemia. Novolin^®R will be used to induce hypoglycemia.
  Interventions: Drug: SAR438544; Drug: insulin
- Glucagon (Active Comparator): Single dose of glucagon given SC under fasting conditions and under induced hypoglycemia. Novolin^®R will be used to induce hypoglycemia.
  Interventions: Drug: r-glucagon; Drug: insulin
- SAR438544 Optional Dose (Experimental): Optional lower, intermediate, or higher dose of SAR438544 given SC under fasting conditions and under induced hypoglycemia. Novolin^®R will be used to induce hypoglycemia.
  Interventions: Drug: SAR438544; Drug: insulin

INTERVENTIONS:
Drug: SAR438544 — Pharmaceutical form:solution
  Route of administration: subcutaneous
  Arms: SAR438544 Optional Dose; SAR438544 dose 1
Drug: r-glucagon — Pharmaceutical form:solution
  Route of administration: subcutaneous
  Other Names: GlucaGen® HypoKit
  Arms: Glucagon
Drug: insulin — Pharmaceutical form:solution
  Route of administration: intravenous
  Other Names: Novolin® R

SUMMARY:
Primary Objective:

To assess the pharmacodynamic response (PD) of a single subcutaneous (SC) dose of SAR438544 versus recombinant glucagon in type 1 diabetes mellitus (T1DM) patients under induced hypoglycemia.

Secondary Objective:

To assess the safety and tolerability and pharmacokinetics (PK) of a single SC dose of SAR438544 versus recombinant glucagon in T1DM patients under induced hypoglycemia.

DETAILED DESCRIPTION:
The total duration of study per patient is up to 8 weeks with 3 to 28 days screening period, 1 day for treatment for both periods and 7 to 14 days wash out between 2 administrations, and 7 days (+/- 1 day) follow-up after last IMP administration.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients, between 18 and 60 years of age, inclusive, with T1DM for at least one year, as defined by the American Diabetes Association (ADA).
* Total (basal+short acting) daily insulin dose of <1.2 U/kg/day.
* Body weight between 50.0 and 110 kg, inclusive, the body mass index (BMI) between 18.5 and 30.0 kg/m^2, inclusive.
* Fasting serum C-peptide <0.3 nmol/L.
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9%).
* Stable insulin regimen for at least 2 months prior to study and self-monitoring of blood glucose before screening visit.
* Certified as otherwise healthy for T1DM by assessment of medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculoskeletal system), unless the Investigator considers any abnormality to be clinically irrelevant and not interfering with the conduct of the study.
* Female subject must use a double contraception method, including a highly effective method of birth control, except if she has undergone sterilization defined as tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and bilateral tubal ligation at least 3 months earlier or is postmenopausal.

The accepted double contraception methods include the use of intrauterine device or hormonal contraception started at least 30 days prior to the screening start and continued for at least 3 months after IMP dosing in addition to one of the following contraceptive options: (1) condom plus spermicide; (2) diaphragm plus spermicide or cervical/vault cap plus spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma follicle-stimulating hormone (FSH) level >30 UI/L in women older than 40 years of age.

* Having given written informed consent prior to undertaking any study-related procedure.
* Not under any administrative or legal supervision.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom, diaphragm or cervical cap, plus spermicide) plus (intra-uterine device or hormonal contraceptive) from the inclusion up to 3 months after the last dosing (except if sterilized).
* Male subject whose partners are pregnant must use during sexual intercourse a condom from the inclusion up to 3 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 3 months after the last dosing.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular (includes ischemia, atrioventricular (AV) block; arrhythmias), pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from T1DM), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent severe headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood loss (>300 mL) within 3 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure (BP), or asymptomatic postural hypotension defined as a decrease in systolic BP ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-HCG] blood test), breast-feeding at screening and before any treatment periods (defined as positive β-HCG urine test).
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis C virus (HCV) Abs, anti-human immunodeficiency virus 1 (HIV1) and anti-HIV2 Abs, and HIV1 Ag.
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol breath test.
* Known hypersensitivity to glucagon, lactose or any other constituent in GlucaGen^® HypoKit and SAR438544 or Novolin^®R and their excipients.
* Any contraindication from the use of glucagon:
* Pheochromocytoma
* Insulinoma and glucagonoma

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Time to reach a smoothed blood glucose of 70 mg/dL after initial administration of investigational medicinal product | Day 1

SECONDARY OUTCOMES:
Assessment of PD parameter: continuous monitoring of blood glucose levels over a period of 6 hours post-dose | Day 1
Assessment of PD parameter: area under plasma concentration of the BG-time curve between IMP dosing and time t (BG-AUC0-t) | Day 1
Assessment of PD parameter: BG-maximum concentration (BG-Cmax) | Day 1
Assessment of PD parameter: BG-time to Cmax (BG-tmax) | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): Cmax | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): tmax | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): tlast | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): terminal half-life | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): area under curve from zero time until the last measurable concentration (AUClast) | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): AUC | Day 1
Assessment of PK parameter (recombinant glucagon and SAR438544): partial AUCs (AUC0-t) | Day 1
Number of patients with adverse events | Day 1 to Day 7 (+/- 1 day)
Time to reach a smoothed blood glucose of 90 mg/dL after initial administration of investigational medicinal product | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi